CLINICAL TRIAL: NCT04201951
Title: Tranexamic Acid for the Prevention of Blood Loss After Vaginal Delivery in a High Risk Pregnancy: A Double Blind Randomized Controlled Trial
Brief Title: Tranexamic Acid for the Prevention of Blood Loss in High Risk Delivered Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Shahla Alalaf, Professor, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HawlerMU3
Record Dates: First submitted 2019-12-14; First posted 2019-12-17 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Postpartum Hemorrhage; High Risk Pregnancy; Tranexamic Acid; Third-Stage Postpartum Hemorrhage, With Delivery
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Two infusion bags will be prepared and labeled as bag A (experimental group) containing 1 g/10mL Tranexamic acid diluted with 20mL of 5% glucose water, and bag B (placebo group) containing 30 mL of 5% glucose water. Providers and patients will be blinded to the contents of the bags until the end of the study. TA or placebo will be administered intravenously immediately after the delivery of the fetus.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All providers and delivered women will be blinded for the content of the bags which will be applied for women randomly
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic group (Active Comparator): Group A will receive 1gm Tranexamic acide diluted in 20 ML 5% glucose water
  Interventions: Drug: Tranexamic acid injection; Other: Glucose water 5%
- Placebo group (Placebo Comparator): Group B will receive 30ML 5% glucose water
  Interventions: Drug: Tranexamic acid injection; Other: Glucose water 5%

INTERVENTIONS:
Drug: Tranexamic acid injection — Participant in group A will receive 2 ampules of 5 milliliters (mL) Tranexamic acid applied to 20 mL of 5% glucose water slowly intravenously immediately after the delivery of the fetus
  Other Names: TRENAXA 500 mg, MACLEODS PHARMACEUTICALS LTD.India
Other: Glucose water 5% — Group B will receive 30 mL of 5% glucose water slowly intravenously immediately after the delivery of the fetus
  Other Names: Glucose B.Braun 50 mg/mL

SUMMARY:
Postpartum hemorrhage and its complications are very well known causes for maternal mortality .Uterine atony is the most common cause for postpartum hemorrhage

DETAILED DESCRIPTION:
Postpartum hemorrhage and its complications are very well known causes for maternal mortality and morbidity especially in developing countries. World Health Organization Recommendations for Active Management of the Third Stage of Labor (AMTSL), on 2012 included the use of uterotonics for the prevention of postpartum hemorrhage (PPH) during the third stage of labor for all births. Tranexamic acid (TA) is antifibrinolytic agent used to decrease blood loss in surgery and health conditions associated with increased bleeding.

A Cochrane Systematic Review from the best available evidence to determine whether TA is effective and safe for preventing PPH in comparison to placebo or no treatment the review concluded that TA (in addition to uterotonic medications) decreases blood loss postpartum and prevents PPH and blood transfusions following vaginal birth and abdominal delivery in women at low risk of PPH based on studies of mixed quality. There was insufficient evidence to draw conclusions about serious side effects and the effects of TA on venous thromboembolic events and mortality beside its use in high-risk women was not investigated on

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year.
* Planed vaginal delivery
* Grand multiparity
* Twin pregnancy
* Polyhydramnios
* Previous history of PPH
* Macrosomic baby
* Prolonged labour
* HELLP syndrome
* Using of low-molecular weight heparin and Asprin during pregnancy.
* Vaginal birth after Cesarean section

Exclusion Criteria:

* Intrauterine death.
* History of thromboembolic disease
* Current or previous history of heart disease ,renal and liver disorders
* History of seizure or epilepsy
* Placenta previa
* Placental abruptio

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
The amount of vaginal blood loss in the third and fourth stages (the fourth begins with delivery of the placenta and ends 2 hours after delivery) | From the time of injection and up to 2 hours after delivery
  The volume of blood loss vaginally will be measured by weighing a specially prepared pad applied beneath the delivered women buttocks before the delivery of the fetus. An electronic scale will be used to weigh the pads before and after 2 hours of the delivery. The quantity of blood (ml) will be = (weight of used materials - weight of materials prior to use)

SECONDARY OUTCOMES:
Number of participant with Post Partum Hemorrhage | up to 2 hours after delivery
  Vaginal blood loss of more than 500 mL
Number of participant with severe postpartum hemorrhage | up to 2 hours after delivery
  Vaginal blood loss ≥1000mL
Number of participant who will need additional uterotonic drugs to control blood loss | up to 2 hours after delivery
  Methyl Ergometrine 0.2 mL, 20 IU oxytocin , and/or 800 misoprostol rectally
the mean length of third stage of labor in both groups | up to 30 minutes
  time from injection of the intervention and placebo group till the delivery of placenta

CONTACTS AND LOCATIONS:
Overall Officials: Shahla K. Alalaf, professor, Principal Investigator — Hawler Medical University; Sazgar A. Rashid, FIBOG, Study Chair — Ministery of Health; Chro S. Hassan, MBChB, Study Chair — Kurdistan Board for Medical Speciality
Locations (2):
- Iraq (2):
  - Kurdistan Board for Medical speciality, Erbil, Kurdistan Region
  - Maternity Teaching Hospital, Erbil, Kurdistan Region